CLINICAL TRIAL: NCT06079593
Title: GaslEss Macular Hole Surgery (GEM): a Feasibility Study
Brief Title: GaslEss Macular Hole Surgery
Acronym: GEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 204994
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Macular Holes
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Images will be graded in a masked fashion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gasless Surgery (Experimental)
  Interventions: Procedure: Gasless Macular hole surgery
- Standard surgery with gas tamponade (Active Comparator)
  Interventions: Procedure: Standard Macular hole surgery

INTERVENTIONS:
Procedure: Gasless Macular hole surgery — Pars plana vitrectomy to treat full thickness macular hole, with internal limiting membrane flap and ophthalmic viscosurgical device covering
  Arms: Gasless Surgery
Procedure: Standard Macular hole surgery — Pars plana vitrectomy to treat full thickness macular hole, with internal limiting membrane peel, and C2F6 tamponade
  Arms: Standard surgery with gas tamponade

SUMMARY:
Macular holes are a hole in the centre of the retina, the light-sensing layer in the back of the eye. They cause a central 'blind spot' in the vision, which can be very disabling for patients. Standard surgery involves injecting a large gas bubble inside the eye. This takes 4-8 weeks to leave the eye. During this time vision is greatly reduced in the eye. This limits patients' ability to drive and work. Gas causes clouding of the natural lens in the eye (cataract). The gas can also raise pressure inside the eye, causing pain and sometimes loss of vision. Patients cannot fly or have certain medicines until the gas absorbs.

Critically, most patients position face down for 50 minutes out of every hour for a week after surgery. This is to float the gas bubble onto the macula. Head positioning is particularly difficult. It very often causes pain in the neck, back, arms and legs. Rarely, blood clots can form in the legs and be life-threatening if they dislodge and travel to the lungs. Head positioning also places a large burden on those caring for the patient.

The gases are 'greenhouse' gases and cause damage to the environment, for about 3,200 years.

This study looks at a new surgical technique for treating macular holes. The new technique aims to make patients' recovery from surgery easier, and safer.

The purpose of this study therefore is to compare two treatments:

* Standard macular hole surgery with gas tamponade
* Novel macular hole surgery without tamponade Gathering feasibility data to inform a future fully powered trial

DETAILED DESCRIPTION:
The investigators are testing a new surgical technique, that does not use the gas bubble and face down positioning. Instead, a licensed surgical gel and thin flap of retinal tissue seal the macular hole. Early small studies suggest the new technique is safe and works as well as standard surgery.

The investigators will invite 60 people with macular hole to take part in the study. Half will be randomly allocated to the new technique and half to standard surgery. All participants will return at regular intervals after surgery for review. The investigators will test their vision, examine their eyes, and ask participants to complete questionnaires about their treatment and vision.

The investigators aim to examine if the technique appears safe and works well at closing macular holes. It will also inform if a larger clinical trial is possible.

ELIGIBILITY:
Inclusion Criteria:

* Requiring PPV to treat idiopathic (primary) FTMH.
* 18 years or older
* ETDRS BCVA letter score of 1 or better in the study eye
* Able to provide written informed consent

Exclusion Criteria:

General:

* Hypersensitivity to hyaluronate or other components of Healon Pro® viscoelastic
* Any major illness or major surgical procedure within 4 weeks
* Any other condition that, in the opinion of the investigator, would prevent the participant from granting informed consent or complying with the protocol

Study eye

* Previous vitreoretinal surgery, retinopexy, open-globe injury, or endophthalmitis
* Presence of fibrotic retinal proliferation or central epiretinal membrane (within 1 disc diameter of the fovea)
* Aphakia
* Current or former myopia greater than 6 dioptres
* Current or previous posterior uveitis or choroiditis
* Presence of other ocular co-morbidity that, in the opinion of the investigator, is likely to impair BCVA postoperatively or affect FTMH closure
* Current ocular or periocular infection, other than mild or moderate blepharitis
* Lens or media opacity that preclude adequate retinal assessment and imaging

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Screen failure | 36 months
  Proportion of those screened who are randomised
Feasibility: Recruitment rate | 36 months
  Recruitment rate (participants per site per month)
Feasibility: Participant retention | 6 months
  Proportion reaching month 6 milestone visit
Feasibility: Cross-over | 36 months
  Proportion converting to standard vitrectomy with gas, due to inability to seal the FTMH, or detection of peripheral retinal breaks

SECONDARY OUTCOMES:
Efficacy Outcomes: Early Treatment Diabetic Retinopathy Study (ETDRS) best-corrected visual acuity (BCVA) | 6 months
  Mean change from baseline
Efficacy Outcomes: Surgical success | 3 months
  Proportion with FTMH closure within 3 months, without further FTMH surgery
Efficacy Outcomes: Area under the BCVA versus time curve (ETDRS letter score) | 6 months
Safety outcomes: Adverse events | 6 months
Safety outcomes: Intra- and post-operative complications | 6 months
Safety outcomes: Development or progression of lens opacity | 6 months
  Within 6 months of vitrectomy (proportion undergoing or listed for cataract surgery and mean change in Lens Opacities Classification System 2 [LOCS2] grading)
Patient reported outcomes measures: Participant acceptability of the intervention | 6 months
  Assessed by the Macular Disease Treatment Satisfaction Questionnaire (MacTSQ; composite score)
Patient reported outcomes measures: National Eye Institute 25-Item Visual Function Questionnaire (NEI VFQ25; composite score) | 6 months
Patient reported outcomes measures: Qualitative analysis | 6 months
  Analysis of participant feedback

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Jackson, PhD, FRCOphth, Principal Investigator — King's College London & King's College Hospital

REFERENCES:
- [Derived] Murphy GSP, Wafa HA, Tarpey M, Wyatt D, Wang Y, Steel DH, Jackson TL. Gas versus GaslEss surgery for full thickness Macular hole (GEM): study protocol for a randomised, assessor-masked, surgical feasibility study. BMJ Open Ophthalmol. 2025 Dec 25;10(1):e002260. doi: 10.1136/bmjophth-2025-002260. PMID 41448786